CLINICAL TRIAL: NCT03492502
Title: Autologous Fecal Microbiota Transplantation for Patients With Acute Graft-versus-Host Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Haggai Bar-Yoseph MD, Principal investigator, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rambam207
Record Dates: First submitted 2018-03-22; First posted 2018-04-10 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Fecal Microbiota Transplantation in Graft vs. Host Disease
Keywords: Fecal microbiota transplantation; allogeneic stem cell transplantation; microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allo-SCT patients with GI related GVHD (Experimental): Allo-SCT patients above 18 years of age with acute steroid-resistant GI-related GVHD grade III-IV.
  The diagnosis of GVHD will be made on clinical grounds (in line with the major associations' recommendations) - the appearance of characteristic mucoid diarrhea within 100 days after Allo-SCT, with or without associated skin/liver involvement. In cases of atypical presentation - we will recommend biopsy or endoscopy for diagnosis. Patients suspected to have Clostridium difficille associated diarrhea will be tested for toxin (CDT).
  Steroid-resistant GI-related GVHD will be defined as lack of improvement (same stage) or worsening of GI symptoms after 7 days of steroid therapy (≥ 2 ml/kg of IV methylprednisolone).
  Interventions: Biological: Autologous Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Autologous Fecal Microbiota Transplantation — Consenting allo- SCT patients with acute steroid-resistant GI-related GVHD grade III-IV will receive autologous FMT by nasogastric tube. Standardized stool suspension will be given once a day for two consecutive days.In order to prevent aspiration, patients will be kept in a 45ᵒ upright position for four hours. Participants will fast the night before and be treated with proton pump inhibitors prior to each FMT.
  In cases where complete response was not obtained within 7 days after autologous FMT, patients may be eligible for another trail of autologous FMT or to switch to other pharmacological interventions. Stool samples will be collected before and after the intervention for microbial analyses.

SUMMARY:
This study aims to assess the safety and efficacy of autologous fecal microbiota transplantation (FMT) in gastrointestinal (GI) related graft-versus-host disease (GVHD). Stool for FMT will be prepared from pre-allogeneic stem cell transplantation (Allo-SCT) period. This strategy might offer a novel and safe therapeutic approach for these patients, who suffer from high disease related morbidity and mortality and are refractory to multiple treatments.

DETAILED DESCRIPTION:
All candidates for Allo-SCT at BMT unit in RHCC will be screened for study inclusion and exclusion criteria. Seven to fourteen days prior to Allo-SCT (before initiation of SCT related antimicrobials), all consenting patients will supply stool sample (first stool sample), which will serve as the autologous FMT sample, and clinical data will be collected. Patients who will develop GI related GVHD will be asked to supply another stool sample 7±2 days after the appearance of GVHD related symptoms (second stool sample). Clinical and laboratory data will be collected. Another stool sample will be collected 7-14 following autologous FMT (third stool sample), and clinical data and outcome will be documented. Day 1 of the study will be defined as day of Allo-SCT, and follow up period is 6 months. Complementary data will be collected from the electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Allo-SCT patients above 18 years of age with acute steroid-resistant GI-related GVHD grade III-IV.

Exclusion Criteria:

* Prior inclusion to an interventional study
* Pregnant or lactating women
* Previous Allo-SCT
* Known multi-drug resistance carriage prior to stool collection
* Severe colitis of any etiology or a history of inflammatory bowel disease (IBD)
* Uncontrolled infection (hemodynamic instability, ongoing fever or bacteremia within 3 days after antibiotics administration)
* Active GI bleeding
* Absolute neutrophil count < 500 cells/microL
* Patients who cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Development of severe adverse events (SAEs) related to autologous FMT | 7 days
  Development of SAEs related to autologous FMT within 7 days after the intervention. SAEs include mortality, bacteremia, and radiological-proven aspiration pneumonia requiring mechanical ventilation.

SECONDARY OUTCOMES:
Complete or partial response of GI-related GVHD after each FMT | 90 days
  Patients will be evaluated 90 days following FMT for symptoms severity and response. Response is defined as:
  1. Complete response - resolution of all GI symptoms
  2. Partial response - decrease of severity of GI-related GVHD by at least one stage or ability to taper steroids to <0.5 mg/kg
  3. No response - progression of symptoms or no change in GI symptoms
Non-severe adverse events (AE) | 7 days
  Non-severe adverse events including dyspepsia, abdominal pain, nausea, vomiting, diarrhea, constipation, fever, or aspiration not requiring mechanical ventilation. Each AE will be graded.
Mortality | 90 days
Change in microbiota composition after each FMT | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel